CLINICAL TRIAL: NCT00815256
Title: The Safety and Effectiveness of Collagen Cross Linking With Riboflavin and Ultraviolet-A Light in Progressive Mild and Moderate Grades of Keratoconus.
Brief Title: Safety and Effectiveness of Collagen Cross Linking in Progressive Mild and Moderate Keratoconus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Patricia Cabral Zacharias Serapicos, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1970/07
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-11

CONDITIONS: Cornea Degeneration; Progressive Keratoconus
Keywords: Cornea degeneration; keratoconus; collagen cross linking; CXL; Riboflavin
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cross linking (CXL) (Experimental): Patients with progressive mild and moderate grades of ketatoconus are randomized and allocated to this group and submitted to the treatment with riboflavin and ultraviolet -A light. They do not match any of the exclusion criterion: pregnancy, corneal thickness less than 400 μm, history of corneal surgery, herpes ocular infection, other corneal disease or scarring, chemical injuries and riboflavin allergy.
  Interventions: Procedure: Collagen Cross Linking with Riboflavin and UVA light

INTERVENTIONS:
Procedure: Collagen Cross Linking with Riboflavin and UVA light — The patients randomized and allocated to this group are submitted to the treatment with riboflavin and ultraviolet -A light, if they do not match any of the exclusion criterion. The treatment is done as follows:after topical anesthesia, the epithelial tissue was removed in a 8.0mm diameter area of the central cornea, the 0,1% riboflavin solution were applied every 2 min, for 30 min followed by cornea irradiation with UVA light with a wavelength of 370 nm and an irradiance of 3 mW/cm2. During the irradiation, drops of the riboflavin solution were continuously applied onto the cornea every 5 min. After the procedure, a therapeutic contact lens and antibiotic eye ointment are applied onto the cornea for a week. We see the patient in the next day.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of collagen cross linking (CXL) in reducing progression of mild and moderate progressive keratoconus.

DETAILED DESCRIPTION:
Keratoconus is a corneal degeneration characterized by bilateral conical protusion and corneal thinning. The course of the disease varies from slight irregular astigmatism to severe visual impairment due to increasing protrusion and subepithelial scarring. There is no treatment available that can stop keratoconus progression. Thus, because of its progressive nature, keratoconus is the most frequent reason for keratoplasty worldwide in the past 3 decades.

The collagen crosslinking (CXL) technique using riboflavin and ultraviolet - A (UVA) light was recently developed to counteract the progressive corneal thinning, and thus the progression of keratoconus. With crosslinking, additional covalent binding between collagen molecules can be achieved, which stabilizes the collagen scaffold and enhances corneal resistance.

Prospective longitudinal randomized case-control study including progressive keratoconus cases is addressed to evaluate the effectiveness of collagen cross linking (CXL) in reducing progression of mild and moderate progressive keratoconus. Progression is based on increase in the cone apex keratometry of - 0,75 D, alteration of - 0,75 D in the spherical equivalent or increase of the anterior chamber depth on Pentacan, in a period of at least six months. All patients must be between 15 and 40 year old and are randomized and allocated in the treated or the control groups. Complete exam before and after exam included best corrected visual acuity, refraction, IOP, fundoscopy, imaging exams such as corneal computerized topographic, pentacan, orbscan, ultrasound pachymetry, esthesiometry, endothelial cell count, HRT II system confocal microscopy, optic coherence tomography (VISANTE), ORA , optic coherence tomography (Stratus OCT) and dynamic contour tonometry . All the exams are repeated 1, 3, 6 and 12 months after the procedure. The cross linking is performed as follows: after topical anesthesia, the epithelial tissue is removed in a 8.0mm diameter area of the central cornea, the 0,1% riboflavin solution is applied every 2 min, for 30 min followed by cornea irradiation with UVA light with a wavelength of 370 nm and an irradiance of 3 mW/cm2. During the irradiation, drops of the riboflavin solution is continuously applied onto the cornea every 5 min.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus patients, with progression of the disease, based on an increase in the cone apex keratometry of - 0,75 D, alteration of - 0,75 D in the spherical equivalent or increase of the anterior chamber depth on pentacan, in a period of at least six months.

Exclusion Criteria:

* pregnancy, corneal thickness less than 400 μm, history of corneal surgery, herpes ocular infection, other corneal disease or scarring, chemical injuries and riboflavin allergy

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Stop progression of keratoconus in cornea imaging exams | 1, 3, 6 and 12 months

SECONDARY OUTCOMES:
Increase in the collagen fibrils density in the confocal microscopy; sensitivity in the esthesiometry; Keratometry (stabilizes or reduces) in the topography; anterior chamber depth on pentacan; etc | 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Denise D Freitas, Professor, Study Chair — Ophthalmology Department Chair
Locations (1):
- Department of Ophthalmology, Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Raiskup-Wolf F, Hoyer A, Spoerl E, Pillunat LE. Collagen crosslinking with riboflavin and ultraviolet-A light in keratoconus: long-term results. J Cataract Refract Surg. 2008 May;34(5):796-801. doi: 10.1016/j.jcrs.2007.12.039. PMID 18471635